CLINICAL TRIAL: NCT00084747
Title: Phase I/II Trial of Autologous Peripheral Blood Progenitor Cell Transplantation With VELCADE Maintenance as Treatment for Intermediate- and Advanced-Stage Multiple Myeloma
Brief Title: Adjuvant Bortezomib Maintenance Therapy After Autologous Peripheral Stem Cell Transplantation in Treating Patients With Intermediate or Advanced Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000365583; UCLA-0306106; MILLENNIUM-MM2003
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2016-02

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib (Experimental)
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Giving bortezomib as maintenance therapy after autologous stem cell transplantation may kill more cancer cells and prolong remission.

PURPOSE: This phase I/II trial is studying the side effects and best dose of adjuvant bortezomib as maintenance therapy and to see how well it works in treating patients who have undergone stem cell transplantation for intermediate or advanced multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response rate, as defined by resolution of bone marrow plasmacytosis and monoclonal paraproteinemia, in the first year after autologous peripheral blood stem cell transplantation in patients with intermediate or advanced multiple myeloma treated with adjuvant bortezomib.
* Compare progression-free survival of patients treated with adjuvant bortezomib with historical controls treated with autologous transplantation alone.
* Determine the toxicity of this drug in these patients (phase I).

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive bortezomib IV on days 1, 8, and 15. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intermediate or advanced multiple myeloma meeting criteria for at least 1 2 following:
* Intermediate- to high-M-component production rates (immunoglobulin [Ig]G > 5 g/dL or immunoglobulin A (IgA) > 3 g/dL or urine M component > 4 g/24 hours)
* More than one osteolytic bone lesion or radiographic evidence of diffuse osteoporosis
* β-2 microglobulin > 3
* Nonsecretory myeloma if bone marrow plasmacytosis is greater than 30%
* Must have undergone autologous peripheral blood stem cell transplantation within the past 3-4 months
* Age 18 to 69 years old
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 30,000/mm^3
* serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) ≤ 300 IU
* Bilirubin ≤ 2 mg/dL
* Creatinine ≤ 2.0 mg/dL
* Creatinine clearance ≥ 30 mL/min
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion Criteria:

* concurrent major cardiac disease that would preclude study participation
* concurrent major pulmonary disease that would preclude study participation
* pregnant or nursing
* peripheral neuropathy ≥ grade 2
* history of hypersensitivity to bortezomib, boron, or mannitol
* concurrent major gastrointestinal or bladder disease that would preclude study participation
* concurrent major neurologic or psychiatric disease that would preclude study participation
* dementia or significantly altered mental status that would preclude giving informed consent
* prior interferon post-transplantation
* prior thalidomide post-transplantation
* prior chemotherapy post-transplantation
* prior radiotherapy post-transplantation
* prior investigational therapy post-transplantation
* prior bortezomib
* prior therapy for myeloma post-transplantation
* other concurrent anti-myeloma therapy
* other concurrent investigational therapy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary J. Schiller, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Schiller GJ, Sohn JP, Malone P, et al.: Phase I/II trial of bortezomib maintenance following autologous peripheral blood progenitor cell transplantation as treatment for intermediate- and advanced-stage multiple myeloma. [Abstract] Biol Blood Marrow Transplant 13 (2 Suppl 1): A-153, 57, 2007.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib: bortezomib administration beginning 3-4 month after the day of transplantation after resolution of bone marrow transplant toxicities
Period: Overall Study
Arm/Group | Bortezomib
Started | 30
Completed | 17
Not Completed | 13
Not completed — Relapsed | 8
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Disease Progression: The day when bone marrow recurrence and/or new lytic bone marrow lesions on radiograph and/or progressive M-component paraprotein (~ 25% increase) were detected. Paraprotein progression will be confirmed labs on the consecutive month.
Time Frame: signed consent to progression or end of trial. Up to 5 years.
Measure: Median (Full Range); unit: months
Groups:
- Bortezomib: autologous peripheral blood progenitor cell transplantation with bortezomib maintenance as treatment for intermediate-and advanced-stage multiple myeloma
Arm/Group | Bortezomib
Number analyzed (Participants) | 30
months | 29 [18 to 45]

2. Secondary Outcome: Overall Survival
Time Frame: up to 5 years from time of consent
Measure: Median (Full Range); unit: months
Groups:
- Bortezomib: bortezomib
Arm/Group | Bortezomib
Number analyzed (Participants) | 30
months | 55 [16 to 86]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from the time subject signed consent until 30 days post last treatment up to 2 years.
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=30)
Nausea/Dehydration (General disorders) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=30)
Fatigue (General disorders) | 19 (19)
Fever (Infections and infestations) | 1 (1)
Anorexia (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
nausea/vomiting (General disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Infections and infestations) | 4 (4)
Upper Respiratory Infection (Infections and infestations) | 2 (2)
Neuropathy (General disorders) | 11 (11)
Pain (General disorders) | 17 (17)
Peripheral Edema (General disorders) | 1 (1)
Herpes Zoster Reactivation (Immune system disorders) | 7 (7)
Rash (General disorders) | 2 (2)
Neutrophils (General disorders) | 6 (6)
Platelets (General disorders) | 10 (10)
Transaminits 2/2 Hep A from contaminated food (Infections and infestations) | 1 (1) — not related
Right extremity swelling, with no DVT (General disorders) | 1 (1) — not drug related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No